CLINICAL TRIAL: NCT01728025
Title: Long Term Prophylactic Therapy of Congenital Long QT Syndrome Type III (LQT3) With Ranolazine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-12-SV-0363-10-CTIL
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Long QT Syndrome Type 3
Keywords: Long QT syndrome; Ranolazine
MeSH Terms: conditions — Long QT syndrome type 3; Long QT Syndrome | interventions — Ranolazine

ARMS (1):
- Ranolazine (Experimental): Ranolazine 500-1000 mg twice a day as tolerated
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine
  Other Names: Ranexa

SUMMARY:
The purpose of this study is to determine whether ranolazine will reduce the risk of arrhythmic events in patients with long QT syndrome type 3.

ELIGIBILITY:
Inclusion Criteria:

* Long QT patients with genetic confirmation of carrier-status for the D1790G mutation in the SCN5A gene
* Corrected QT interval > 460 msec

Exclusion Criteria:

* Need for therapy with medications that are potent or moderately potent CYP3A inhibitors (such as ketoconazole, diltiazem, verapamil, macrolide antibiotics or HIV protease inhibitors)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with syncope and/or documented ventricular arrhythmia | 5 years

SECONDARY OUTCOMES:
Change in corrected QT interval | within 30 days of initiation of Ranolazine treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Moss AJ, Zareba W, Schwarz KQ, Rosero S, McNitt S, Robinson JL. Ranolazine shortens repolarization in patients with sustained inward sodium current due to type-3 long-QT syndrome. J Cardiovasc Electrophysiol. 2008 Dec;19(12):1289-93. doi: 10.1111/j.1540-8167.2008.01246.x. Epub 2008 Jul 25. PMID 18662191
- [Background] Lindegger N, Hagen BM, Marks AR, Lederer WJ, Kass RS. Diastolic transient inward current in long QT syndrome type 3 is caused by Ca2+ overload and inhibited by ranolazine. J Mol Cell Cardiol. 2009 Aug;47(2):326-34. doi: 10.1016/j.yjmcc.2009.04.003. Epub 2009 Apr 14. PMID 19371746
- [Derived] Chorin E, Hu D, Antzelevitch C, Hochstadt A, Belardinelli L, Zeltser D, Barajas-Martinez H, Rozovski U, Rosso R, Adler A, Benhorin J, Viskin S. Ranolazine for Congenital Long-QT Syndrome Type III: Experimental and Long-Term Clinical Data. Circ Arrhythm Electrophysiol. 2016 Oct;9(10):e004370. doi: 10.1161/CIRCEP.116.004370. PMID 27733495